CLINICAL TRIAL: NCT01527318
Title: The Effect of Fibrate Therapy in Two Patients With Neutral Lipid Storage Disease With Myopathy (NLSDM)
Acronym: NLSDM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEC 11-3-013
Record Dates: First submitted 2012-01-16; First posted 2012-02-07 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Neutral Lipid Storage Disease
Keywords: NLSDM; Lipid accumulation
MeSH Terms: conditions — Chanarin-Dorfman Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fibrate Treatment (Experimental): Patients will be treated during 28 weeks with a fibrate to assess the effects of PPAR activation on the NLSDM disease.
  Interventions: Drug: Fibrate treatment

INTERVENTIONS:
Drug: Fibrate treatment — Patients will receive a dosage of 400mg Bezafibrate every day during 28 weeks

SUMMARY:
Neutral Lipid Storage Disease With Myopath (NLSDM) is a disease caused by a defect in the PNPLA2 gene encoding ATGL. Patients with NLSDM accumulate triglycerides and exhibit muscle weakness, cardiac failure and hepatosteatosis. Most of these patients die at young age due to cardiac failure. Not much is known about the underlying mechanisms, though recently it was discovered that PPAR activation in ATGL-/- mice was impaired leading to decreased mitochondrial function, lipid accumulation and cardiac failure resulting in death at young age. Activation of PPARs, by treatment with fibrates rescued the phenotype and reduced mortality rates in these mice. These findings may have a major impact for patients with NLSDM if these results can be translated to humans. Therefore, the investigators would like to evaluate the beneficial effects of fibrate treatment on muscle mitochondrial and cardiac function in patients with NLSDM.

Patients will be treated with fibrates during a period of 28 weeks. Baseline measurements will be performed prior to the study and after treatment. Cardiac and muscular lipid accumulation, cardiac function, mitochondrial function and insulin sensitivity will be assessed during these baseline measurements.

ELIGIBILITY:
Inclusion Criteria:

* suffering from NLSDM

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
mitochondrial function | 28 weeks
  mitochondrial function will be measured in vivo with 1H-MRS by pCr-recovery and ex vivo by high resolution respirometry.
lipid accumulation | 28 weeks
  Lipid accumulation will be measured both by 1H-MRS as CH/H2O ratio's in the Tibialis anterior muscle, as well as quantified from skeletal muscle biopsy with ORO from the vastus lateralis muscle.
Cardiac function | 28 weeks
  Cardiac function will be measured with ultrasound and be assessed by 2 blinded cardiologists.

SECONDARY OUTCOMES:
Insulin sensitivity | 28 weeks
  This will be assessed by an euglycemic hyperinsulenemic clamp and whole body isulin sensitivity will be expressed with the M-value.

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

REFERENCES:
- [Background] Haemmerle G, Moustafa T, Woelkart G, Buttner S, Schmidt A, van de Weijer T, Hesselink M, Jaeger D, Kienesberger PC, Zierler K, Schreiber R, Eichmann T, Kolb D, Kotzbeck P, Schweiger M, Kumari M, Eder S, Schoiswohl G, Wongsiriroj N, Pollak NM, Radner FP, Preiss-Landl K, Kolbe T, Rulicke T, Pieske B, Trauner M, Lass A, Zimmermann R, Hoefler G, Cinti S, Kershaw EE, Schrauwen P, Madeo F, Mayer B, Zechner R. ATGL-mediated fat catabolism regulates cardiac mitochondrial function via PPAR-alpha and PGC-1. Nat Med. 2011 Aug 21;17(9):1076-85. doi: 10.1038/nm.2439. PMID 21857651